CLINICAL TRIAL: NCT00067535
Title: Potential Interactions Between IV Cocaine and RPR 102681
Brief Title: Assessment of Potential Interactions Between Cocaine and RPR 102681 - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NIDA-CPU-0003-1
Record Dates: First submitted 2003-08-21; First posted 2003-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-02

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Cocaine-Related Disorders

SUMMARY:
The purpose of this study is to assess Potential Interactions Between iv Cocaine and RPR 102681

DETAILED DESCRIPTION:
Phase I, Double-Blind, Placebo-Controlled Dose Escalating Assessment of Potential Interactions Between Intravenous Cocaine and RPR 102681

ELIGIBILITY:
Inclusion Criteria:

Includes but is not limited to:

* Non-treatment seekers
* DSM-IV criteria for cocaine abuse or dependence
* Ability to verbalize understanding of consent form and provide written informed consent and verbalize willingness to complete study procedures; be able to comply with protocol requirements

Exclusion Criteria:

Please contact site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response to cocaine and subjective response to cocaine | 3x / 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States